CLINICAL TRIAL: NCT01973582
Title: A Retrospective Cohort Study of Hepatitis B Seroepidemiology Among Young Adults
Brief Title: Hepatitis B Seroepidemiology Among Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201012127RB
Record Dates: First submitted 2013-10-20; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; epidemiology; youth; vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, blood cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Taiwan has launched a successful nationwide neonatal hepatitis B immunization since July 1, 1984. It successfully decreased the incidence of hepatitis B virus infection, the hepatitis B carrier rate as well as liver diseases among children and adolescents. The sexual transmission route is another important way of hepatitis B infection aside from the mother and child vertical infection, especially for youth and adults. Hepatitis B vaccination cohort refers to those who were born after 1986 and received hepatitis B vaccine immunization during newborn period. They are gradually entering into young adults and adolescent age. Among them, there is no empirical evidence to show the actual infection rate and to help implement hepatitis B vaccine booster policy for those who had three seronegative viral markers of hepatitis B. Therefore, the study design is to collect three consecutive years graduate school students school entry health examination data and undergo three hepatitis B viral markers checkup and blood types. The data linkage includes their health checkup data in the freshmen period, Taiwan CDC databank for neonatal hepatitis B immunization records, pregnancy and birth record registry, Taiwan cancer registry and Taiwan death record registry.

DETAILED DESCRIPTION:
This study is aimed to delineate the hepatitis B seroepidemiology among young adults with or without neonatal hepatitis B immunization, among young adults with hepatitis B booster in the university period, among the mothers of hepatitis B vaccination cohort. The results of this study will provide important information to help government implement hepatitis B vaccine booster policy in the adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Young adults 20 to 30 years old.

Exclusion Criteria:

* Refused to undergo blood draw or questionaire.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults 20 to 30 years old.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
serostatus of hepatitis B viral markers | One year

CONTACTS AND LOCATIONS:
Overall Officials: Chyi-Feng Jan, MD, MSc, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Jan CF, Huang KC, Chien YC, Greydanus DE, Davies HD, Chiu TY, Huang LM, Chen CJ, Chen DS. Determination of immune memory to hepatitis B vaccination through early booster response in college students. Hepatology. 2010 May;51(5):1547-54. doi: 10.1002/hep.23543. PMID 20209603
- [Background] Chien YC, Jan CF, Kuo HS, Chen CJ. Nationwide hepatitis B vaccination program in Taiwan: effectiveness in the 20 years after it was launched. Epidemiol Rev. 2006;28:126-35. doi: 10.1093/epirev/mxj010. Epub 2006 Jun 16. PMID 16782778